CLINICAL TRIAL: NCT05056402
Title: Immunogenicity Non-inferiority Immuno-bridging Study of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine (E.Coli) in Healthy Population Aged 9-17 Years Old vs Aged 18-26 Years Old
Brief Title: An Immuno-bridging Study of a Nonavalent HPV Vaccine (E.Coli) in Healthy Population Aged 9-17 vs Aged 18-26 Years Old
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPV-PRO-012
Record Dates: First submitted 2021-09-13; First posted 2021-09-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Condylomata Acuminata
Keywords: human papillomavirus vaccine; immunogenicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 9-17y (0,6m) (Experimental): Subjects who aged 9-17 years old would receive 2 doses of 270μg/0.5ml Recombinant HPV nonavalent (Types 6/11/16/18/31/33/45/52/58) Vaccine(E.Coli) .
  Interventions: Biological: 2 doses of theRecombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli)
- 9-17y (0,1,6m) (Experimental): Subjects who aged 9-17 years old would receive 3 doses of 270μg/0.5ml Recombinant HPV nonavalent (Types 6/11/16/18/31/33/45/52/58) Vaccine(E.Coli) .
  Interventions: Biological: 3 doses of the Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli)
- 18-26y (0,1,6m) (Experimental): Subjects who aged 18-26 years old would receive 3 doses of 270μg/0.5ml Recombinant HPV nonavalent (Types 6/11/16/18/31/33/45/52/58) Vaccine(E.Coli) .
  Interventions: Biological: 3 doses of the Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli)

INTERVENTIONS:
Biological: 3 doses of the Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli) — Three doses administered intramuscularly at 0, 1 and 6 month.
  Arms: 18-26y (0,1,6m); 9-17y (0,1,6m)
Biological: 2 doses of theRecombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli) — Two doses administered intramuscularly at 0 and 6 month.
  Arms: 9-17y (0,6m)

SUMMARY:
This is a open label clinical trial to evaluate the safety and immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58)Vaccine(E.Coli) manufactured by Xiamen Innovax Biotech CO., Ltd., in healthy population aged 9-17 years old in comparison with aged 18-26.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female between and including 9-26 years of age, or male between and including 9-17 years of age at the first vaccination;
2. Subject (and their legal guardian) is able to understand and comply with the requirements of the protocol(e.g. biological specimen collection, completion of the diary cards, return for follow-up visits), and written informed consent must be obtained from the subject prior to enrollment;
3. Adolescent female subject who agrees to practice effective contraception within 8 months after the first vaccination or has undergone tubal ligation,subtotal hysterectomy for benign lesion, ovarian benign tumor resection;
4. No previous history of sexually transmitted diseases (including syphilis, gonorrhea, chancroid, venereal lymphogranuloma, groin granuloma, etc.);
5. Male, or female without previous history of abnormal cervical screening results or cervical intraepithelial neoplasia (CIN);

Exclusion Criteria:

1. Axillary temperature > 37.2℃;
2. Adolescent female subject who has a positive urine pregnancy test, or is pregnant or breastfeeding;
3. Subject has used of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of study vaccine or plans to use during the study period , or has participated in another clinical research in the past two years, or plans to participate in another research during the study period;
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs or systemic corticosteroids (Except intranasal steroid, the use of low dose topical, ophthalmic and inhaled steroid preparations will be permitted.) within 6 months prior to vaccination.
5. Administration of immunoglobulin and/or blood products within 3 months prior to vaccination or planned to use them within 7 months after the first dose.
6. Administration of inactivated vaccine within 14 days prior to vaccination or live vaccine within 21 days;
7. Fever (Axillary temperature ≥38.0℃) 3 days prior to vaccination or system administration of antibiotics or antiviral agents within 5 days, or medicines containing antipyretic ingredients within 24 hours prior to vaccination;
8. Subject has received other HPV vaccines or participated in clinical research related to HPV or cervical cancer previously;
9. Subject has severe immunodeficiency disease, severe primary disease of important viscera, cancer and autoimmune disease (including systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy due to any condition, and other immunological diseases that investigators believe may influence the immune response).
10. History of severe allergy (e.g., anaphylaxis, generalized urticaria, dyspnea, angioedema, and other significant reaction) to any previous vaccination, or be allergic to any of the components of the study vaccines.
11. Asthma, which has been unstable for the past two years and requires emergency treatment, hospitalization, oral or intravenous corticosteroids;
12. Subject has serious medical disorders;
13. Self-report (subject and their legal guardian) coagulation disorders or abnormal coagulation function;
14. Epilepsy, excluding febrile epilepsy under 2 years of age, alcoholic epilepsy 3 years prior to abstinence or simple epilepsy that does not require treatment in the past 3 years;
15. Medical, psychological, social conditions, occupation or other factors, which considered by the investigator that may influence the conduct of the clinical study.

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1382 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity1: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific antibody levels at Months 7 in the population aged 9-26 years old receiving 3 doses of the nonavalent vaccine | 7 months after the first dose
  To determine whether the immune responses (antibodies to HPV-6, 11, 16, 18, 31, 33, 45, 52, and 58) at month 7 (one month after the final dose) in the population aged 9-17 years receiving 3 doses of the nonavalent vaccine are noninferior to those in women aged 18-26 years receiving 3 doses of vaccine.

SECONDARY OUTCOMES:
Immunogenicity2: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific antibody levels at Months 7 in the population aged 9-14 years old receiving 2 doses of the nonavalent vaccine | 7 months after the first dose
  To determine whether the immune responses (antibodies to HPV-6, 11, 16, 18, 31, 33, 45, 52, and 58) at month 7 (one month after the final dose) in the population aged 9-14 years receiving 2 doses of the nonavalent vaccine are noninferior to those in women aged 18-26 years receiving 3 doses of vaccine.
Immunogenicity3: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific antibody levels at months 18 and 30 in the population aged 9-14 and 15-17 years old receiving 2 doses or 3 doses of the nonavalent vaccine | 30 months after the first dose
  To determine the immune persistence (antibodies to HPV-6, 11, 16, 18, 31, 33, 45, 52, and 58) at months 18 and 30 in the population receiving 2 doses or 3 doses of the nonavalent vaccine
Safety1: Local and systematic adverse events/reactions occurred within 7 days after each vaccination. | During the 7-day period following each vaccination
  Local and systematic adverse events/reactions occurred within 7 days after each vaccination.
Safety2: Adverse events/reactions occurred within 30 days after each vaccination. | Within 30 days (Day 0-30) after any vaccination
  Adverse events/reactions occurred within 30 days after each vaccination.
Safety3: Severe adverse events occurred throughout the study. | Up to 8 month
  Severe adverse events occurred throughout the study. To evaluate number of SAEs between the different arms.
Safety4: Pregnancy and pregnancy outcome. | Up to 8 month
  Pregnancy and pregnancy outcome. To evaluate number of births and terminations between the different arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, master, Study Chair — Xiamen University; Xue-cheng Liu, master, Principal Investigator — Sichuan Provincial Centre for Disease Control and Prevention
Locations (1):
- Sichuan Provincial Centre for Disease Control and Prevention, Chengdu, Sichuan, China